CLINICAL TRIAL: NCT05545553
Title: A Randomized Split Mouth Clinical Trial Comparing Piezosurgery and Conventional Rotary Instruments on Impacted Third Molar Surgery
Brief Title: Piezosurgery and Conventional Rotary Instruments on Third Molar Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Ferit Bayram, Assistant Professor, Marmara University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MUDHF_FB_0001
Record Dates: First submitted 2022-09-09; First posted 2022-09-19 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Impacted Third Molar Tooth
Keywords: Impacted Tooth; Piezo-Electric Surgery; Postoperative Complication
MeSH Terms: conditions — Tooth, Impacted; Postoperative Complications | interventions — Piezosurgery

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Piezosurgery group (Experimental): In the experimental group, a piezosurgery device was used to remove the bone surrounding the impacted third molar.
  Interventions: Device: Piezosurgery
- Conventional group (Active Comparator): In the control group, conventional burs were used to remove the bone surrounding the impacted third molar.
  Interventions: Device: Conventional burs

INTERVENTIONS:
Device: Piezosurgery — Piezosurgery used as an osteotomy device
  Arms: Piezosurgery group
Device: Conventional burs — Conventional burs used as an osteotomy device
  Arms: Conventional group

SUMMARY:
The aim of this study is to compare piezosurgery and conventional surgery in impacted third molar surgery and to determine its effect on postoperative outcomes and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II
* Aged 18-35
* Symmetrical Class 2 Position B according to Winter and Pell-gregory classification
* Asymptomatic lower third molar tooth with the same difficulty according to the Yuasa difficulty index

Exclusion Criteria:

* Individuals who had systemic disease affecting bone or soft tissue metabolism
* Smokers (more than 10 cigarettes a day
* Alcohol dependent
* Systemic disease affecting bone or soft tissue metabolism
* Acute pericoronitis or acute periodontal disease at the time of operation, and used antibiotics due to acute infection

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Change in Oral Health-related Quality of Life | 14 days
  Evaluated by OHIP-14

SECONDARY OUTCOMES:
Change in pain | 7 days
  Postoperative pain was assessed using a Visual Analogue Scale (VAS) ranging from the absence of pain (score 0) to the most severe pain imaginable
Change in Mouth opening | 7 days
  The distance between the mesio-incisal corners of the upper and lower central incisors was measured with the help of a ruler when the mouth opening was at its maximum.
Operation time | Intraoperative
  The total time from the first incision of the operation site to the last suture was measured with the help of a digital stopwatch as the operation time.
Change in facial swelling | 7 days
  With the technique described by Neupert ;
  * Angle of mandible-tragus
  * Angle of mandible-lateral canthus of eye
  * Mandible corner-nose wing
  * Angle of mandible oral-commissures
  * Measurements were made with a tape measure from 5 points, with the mandible corner-pogonion.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University School of Dentistry, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
Time Frame: Data will become available in 1 month and will be available for 2 years

REFERENCES:
- [Background] Rullo R, Addabbo F, Papaccio G, D'Aquino R, Festa VM. Piezoelectric device vs. conventional rotative instruments in impacted third molar surgery: relationships between surgical difficulty and postoperative pain with histological evaluations. J Craniomaxillofac Surg. 2013 Mar;41(2):e33-8. doi: 10.1016/j.jcms.2012.07.007. Epub 2012 Aug 11. PMID 22890087
- [Background] Rosa AL, Carneiro MG, Lavrador MA, Novaes AB Jr. Influence of flap design on periodontal healing of second molars after extraction of impacted mandibular third molars. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2002 Apr;93(4):404-7. doi: 10.1067/moe.2002.122823. PMID 12029279
- [Background] Ren YF, Malmstrom HS. Effectiveness of antibiotic prophylaxis in third molar surgery: a meta-analysis of randomized controlled clinical trials. J Oral Maxillofac Surg. 2007 Oct;65(10):1909-21. doi: 10.1016/j.joms.2007.03.004. PMID 17884515
- [Background] Cho H, David MC, Lynham AJ, Hsu E. Effectiveness of irrigation with chlorhexidine after removal of mandibular third molars: a randomised controlled trial. Br J Oral Maxillofac Surg. 2018 Jan;56(1):54-59. doi: 10.1016/j.bjoms.2017.11.010. Epub 2017 Dec 6. PMID 29223633
- [Background] Piersanti L, Dilorenzo M, Monaco G, Marchetti C. Piezosurgery or conventional rotatory instruments for inferior third molar extractions? J Oral Maxillofac Surg. 2014 Sep;72(9):1647-52. doi: 10.1016/j.joms.2014.04.032. Epub 2014 May 6. PMID 25109581
- [Background] Ge J, Yang C, Zheng JW, He DM, Zheng LY, Hu YK. Four osteotomy methods with piezosurgery to remove complicated mandibular third molars: a retrospective study. J Oral Maxillofac Surg. 2014 Nov;72(11):2126-33. doi: 10.1016/j.joms.2014.05.028. Epub 2014 Jun 14. PMID 25201232
- [Background] Barone A, Marconcini S, Giacomelli L, Rispoli L, Calvo JL, Covani U. A randomized clinical evaluation of ultrasound bone surgery versus traditional rotary instruments in lower third molar extraction. J Oral Maxillofac Surg. 2010 Feb;68(2):330-6. doi: 10.1016/j.joms.2009.03.053. Epub 2010 Jan 15. PMID 20116704
- [Background] Goyal M, Marya K, Jhamb A, Chawla S, Sonoo PR, Singh V, Aggarwal A. Comparative evaluation of surgical outcome after removal of impacted mandibular third molars using a Piezotome or a conventional handpiece: a prospective study. Br J Oral Maxillofac Surg. 2012 Sep;50(6):556-61. doi: 10.1016/j.bjoms.2011.10.010. Epub 2011 Nov 15. PMID 22088359
- [Background] Sortino F, Pedulla E, Masoli V. The piezoelectric and rotatory osteotomy technique in impacted third molar surgery: comparison of postoperative recovery. J Oral Maxillofac Surg. 2008 Dec;66(12):2444-8. doi: 10.1016/j.joms.2008.06.004. PMID 19022121
- [Background] Mantovani E, Arduino PG, Schierano G, Ferrero L, Gallesio G, Mozzati M, Russo A, Scully C, Carossa S. A split-mouth randomized clinical trial to evaluate the performance of piezosurgery compared with traditional technique in lower wisdom tooth removal. J Oral Maxillofac Surg. 2014 Oct;72(10):1890-7. doi: 10.1016/j.joms.2014.05.002. Epub 2014 May 13. PMID 25234524
- [Background] Cicciu M, Stacchi C, Fiorillo L, Cervino G, Troiano G, Vercellotti T, Herford AS, Galindo-Moreno P, Di Lenarda R. Piezoelectric bone surgery for impacted lower third molar extraction compared with conventional rotary instruments: a systematic review, meta-analysis, and trial sequential analysis. Int J Oral Maxillofac Surg. 2021 Jan;50(1):121-131. doi: 10.1016/j.ijom.2020.03.008. Epub 2020 Apr 11. PMID 32284166
- [Derived] Demirci A, Bayram F, Dergin G. Piezosurgery versus conventional rotary surgery for impacted third molars: A randomised, split-mouth, clinical pilot trial. Med Oral Patol Oral Cir Bucal. 2024 Jan 1;29(1):e1-e8. doi: 10.4317/medoral.25929. PMID 37992138